CLINICAL TRIAL: NCT04260191
Title: A Global Phase 1 Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of the Half-life Extended Bispecific T-cell Engager AMG 910 in Subjects With Claudin 18.2-Positive Gastric and Gastroesophageal Junction Adenocarcinoma
Brief Title: Study of AMG 910 in Subjects With CLDN18.2-Positive Gastric and Gastroesophageal Junction Adenocarcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20180292
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Results first posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2023-04

CONDITIONS: Gastric and Gastroesophageal Junction Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: AMG 910 6.5 μg (Experimental): For Cycles 1 and 2, participants received AMG 910 as a short-term intravenous (IV) infusion (approximately 60 minutes) at a dose of 6.5 μg twice a week on Days 1 and 3 of each week in a 28-day cycle. For Cycles 3 to 6, participants received AMG 910 as a short-term IV infusion (approximately 60 minutes) at a dose of 6.5 μg weekly, ie, Days 1, 8, 15 and 22 in a 28-day cycle.
  Interventions: Drug: AMG 910
- Cohort 1b: AMG 910 6.5 μg (Experimental): For Cycle 1 Week 1, participants received AMG 910 as an extended IV (eIV) infusion (approximately 96 hours) at a dose of 6.5 μg. For the remainder of Cycles 1 and 2, participants received AMG 910 as a short-term IV infusion (approximately 60 minutes) at a dose of 6.5 μg twice a week on Days 1 and 3 of each week in a 28-day cycle. For Cycles 3 to 6, participants received AMG 910 as a short-term IV infusion (approximately 60 minutes) at a dose of 6.5 μg weekly, ie, Days 1, 8, 15 and 22 in a 28-day cycle.
  Interventions: Drug: AMG 910
- Cohort 2b: AMG 910 15 μg (Experimental): For Cycle 1 Week 1, participants received AMG 910 as an eIV infusion (approximately 96 hours) at a dose of 15 μg. For the remainder of Cycles 1 and 2, participants received AMG 910 as a short-term IV infusion (approximately 60 minutes) at a dose of 15 μg twice a week on Days 1 and 3 of each week in a 28-day cycle. For Cycles 3 to 6, participants received AMG 910 as a short-term IV infusion (approximately 60 minutes) at a dose of 15 μg weekly, ie, Days 1, 8, 15 and 22 in a 28-day cycle.
  Interventions: Drug: AMG 910

INTERVENTIONS:
Drug: AMG 910 — IV Infusion

SUMMARY:
To evaluate the safety and tolerability of AMG 910 in adult subjects, and to determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D)

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically or cytologically confirmed metastatic or locally advanced unresectable gastric or GEJ adenocarcinoma positive for CLDN18.2.
* Subjects should not be eligible for curative surgery and should have been refractory to or have relapsed after two or more prior lines of standard systemic therapy that included a platinum, a fluoropyrimidine, either a taxane or irinotecan, and an approved vascular endothelial growth factor receptor (VEGFR) antibody/tyrosine kinase inhibitor (TKI) and depending on country-specific standards and approvals.
* For subjects eligible for human epidermal growth factor receptor 2 (HER2) directed therapy, prior systemic therapy should have included a HER2 targeting antibody approved for treatment of gastric cancer.
* Subjects may also be included if the aforementioned therapeutic options were medically not appropriate for them. In these cases, the reason(s) why required prior therapies for gastric cancer were medically not appropriate should be documented in the subject's electronic case report form (eCRF).
* For dose-expansion only: Subjects with at least 1 measurable lesion greater than or equal to 10mm which has not undergone biopsy within 3 months of screening scan. This lesion cannot be biopsied at any time during the study.
* Subjects with stable condition and anti-coagulative therapy ongoing for at least 1 month, no obvious signs and symptoms of bleeding, and coagulation parameters are fulfilled.
* Subjects should be able to use proton pump inhibitors.

Exclusion Criteria:

* Any anticancer therapy or immunotherapy within 4 weeks of start of first dose (14 days for palliative radiation).
* Untreated or symptomatic central nervous system (CNS) metastases, leptomeningeal disease, or spinal cord compression
* Autoimmune disorders requiring chronic systemic steroid therapy or any other form of immunosuppressive therapy while on study, eg, ulcerative colitis, Crohn's disease, or any other gastrointestinal autoimmune disorder causing chronic nausea, vomiting, or diarrhea. Recent or current use of inhaled steroids or physiological substitution in case of adrenal insufficiency is not exclusionary.
* Evidence or history within last 3 months of gastrointestinal inflammatory conditions not associated with the underlying cancer disease including gastrinomas, duodenitis, proven gastric ulcer, duodenal ulcer, pancreatitis, or subjects with recent gastric bleeding. Subjects may be included if the symptomatic/immunosuppressive treatment is discontinued more than 4 weeks prior to the first dose of AMG 910, symptoms have resolved, and gastroscopy does not indicate signs of active disease.
* Subjects with inherited bleeding disorders (eg, Willebrand's disease, hemophilia A and other clotting factor deficiency) and subjects with known heparin-induced thrombocytopenia.
* Subjects requiring non-steroidal anti-inflammatory drugs (NSAIDs) during study treatment. The NSAID(s) should be stopped within 7 days prior to start of treatment.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (20):
- United States (3):
  - City of Hope National Medical Center, Duarte, California
  - University of California at Irvine Medical Center, Orange, California
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
- Landeskrankenhaus Salzburg, Salzburg, Austria
- Institut Gustave Roussy, Villejuif, France
- Germany (4):
  - Universitaetsklinikum Hamburg Eppendorf Onkologisches Zentrum, Hamburg
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum der Universität München Campus Grosshadern, München
  - Klinikum rechts der Isar, München
- Japan (3):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - National Cancer Center Hospital, Chuo-ku, Tokyo
- Amsterdam UMC - location VUmc, Amsterdam, Netherlands
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Hospital Universitari Vall d Hebron, Barcelona, Catalonia, Spain
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 15 participants were enrolled and received AMG 910 at 10 centers in Europe, South Korea, Taiwan and the United States between 29 June 2020 and 02 June 2022.
Groups:
- Cohort 1: AMG 910 6.5 µg: For Cycles 1 and 2, participants received AMG 910 as a short-term intravenous (IV) infusion (approximately 60 minutes) at a dose of 6.5 µg twice a week on Days 1 and 3 of each week in a 28-day cycle. For Cycles 3 to 6, participants received AMG 910 as a short-term IV infusion (approximately 60 minutes) at a dose of 6.5 µg weekly, ie, Days 1, 8, 15 and 22 in a 28-day cycle.
- Cohort 1b: AMG 910 6.5 µg: For Cycle 1 Week 1, participants received AMG 910 as an extended IV (eIV) infusion (approximately 96 hours) at a dose of 6.5 µg. For the remainder of Cycle 1 (from Day 8) and for Cycles 2 to 6, participants received AMG 910 as a short-term IV infusion (approximately 60 minutes) at a dose of 6.5 µg weekly, ie, Days 1, 8, 15 and 22 in a 28-day cycle.
- Cohort 2b: AMG 910 15 µg: For Cycle 1 Week 1, participants received AMG 910 as an eIV infusion (approximately 96 hours) at a dose of 15 µg. For the remainder of Cycle 1 (from Day 8) and for Cycles 2 to 6, participants received AMG 910 as a short-term IV infusion (approximately 60 minutes) at a dose of 15 µg weekly, ie, Days 1, 8, 15 and 22 in a 28-day cycle.
Period: Overall Study
Arm/Group | Cohort 1: AMG 910 6.5 µg | Cohort 1b: AMG 910 6.5 µg | Cohort 2b: AMG 910 15 µg
Started | 6 | 4 | 5
Received AMG 910 | 6 | 4 | 5
Completed | 1 | 0 | 0
Not Completed | 5 | 4 | 5
Not completed — Decision by Sponsor | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 3
Not completed — Death | 4 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All participants that were enrolled and received at least 1 dose of AMG 910.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: AMG 910 6.5 µg | Cohort 1b: AMG 910 6.5 µg | Cohort 2b: AMG 910 15 µg | Total
Number analyzed (Participants) | 6 | 4 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (14.9) | 54.3 (22.9) | 63.6 (10.7) | 57.9 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 4
  Male | 4 | 3 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 3 | 4 | 13
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2 | 4
  Black or African American | 1 | 0 | 0 | 1
  White | 4 | 2 | 2 | 8
  Other | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Dose-Limiting Toxicity (DLT)
Description: All DLTs were graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. DLTs were defined as any AEs at least possibly related to AMG 910 with an onset within the first 28 days following first dose with any of the following:
  * Grade 2 gastric perforation or fistula
  * Grade ≥ 3 non-hematologic AEs including laboratory abnormalities
  * Re-challenge with AMG 910 after treatment interruption due to any stomach toxicity results in at least same stomach toxicity and is of CTCAE grade ≥ 3 or grade 2 and ongoing for more than 3 days despite optimal supportive treatment
  * Grade 4 thrombocytopenia or grade 3 thrombocytopenia with bleeding
  * Grade 4 neutropenia lasting > 28 days
  * Febrile neutropenia of any grade
  * Anemia requiring transfusion per local or international guidelines in the absence of bleeding
  * Grade 5 toxicity
  * Any other toxicity related to AMG 910 considered significant enough to be qualified as DLT in the opinion of the investigator
Time Frame: Day 1 to Day 28
Population: Safety Analysis Set: All participants that were enrolled and received at least 1 dose of AMG 910. Only participants who received study treatment (at least 80% of the planned dose for Cycle 1) and remained on study through the DLT assessment window were considered DLT-evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: AMG 910 6.5 µg | Cohort 1b: AMG 910 6.5 µg | Cohort 2b: AMG 910 15 µg
Number analyzed (Participants) | 4 | 3 | 5
Participants | 2 | 0 | 1

2. Primary Outcome: Number of Participants Who Experienced a Treatment-emergent AE (TEAE)
Description: A TEAE was defined as any adverse event starting on or after the first administration of investigational product, as determined by the flag indicating if the adverse event started prior to the first dose on the Events case report form, and up to and including 30 days after the last investigational product dose date.
  Evaluation of TEAEs included the number of participants with at least 1 TEAE or treatment-related TEAE. Clinically significant changes in vital signs, electrocardiogram (ECG) and clinical laboratory tests were recorded as TEAEs.
Time Frame: Day 1 to 30 days post-last dose; maximum duration was 10.97 months
Population: Safety Analysis Set: All participants that were enrolled and received at least 1 dose of AMG 910.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: AMG 910 6.5 µg | Cohort 1b: AMG 910 6.5 µg | Cohort 2b: AMG 910 15 µg
Number analyzed (Participants) | 6 | 4 | 5
Participants
  TEAEs | 6 | 4 | 5
  Treatment-related TEAEs | 4 | 4 | 5

3. Secondary Outcome: Maximum Serum Concentration (Cmax) of AMG 910
Description: Mean Cmax values for the dosing intervals following short-term IV infusion (Cohort 1) and following extended IV infusions (Cohorts 1b and 2b) for Cycle 1 Week 1, and for short-term IV infusions in subsequent dosing intervals in Cycle 1. The timing of the pharmacokinetic (PK) sampling for Week 1 (Days 1 - 7) was based on hours after the start of the infusion and from Day 8 onwards was based on hours after the end of infusion (EOI). Due to the limited number of samples obtained and early termination of the study, PK data are summarized for Cycle 1 only.
Time Frame: Cycle 1: Days 1-7 at pre-infusion, 1, 2, 4, 24, 48, 72, 96, 120 and 144 hr; Days 8 and 10* at pre-infusion, EOI, 4 and 24 hr post-EOI; Days 15, 17* and 22* at pre-infusion and EOI; Day 24* at pre-infusion, EOI, 2, 4 and 24 hr post-EOI (*=Cohort 1 only)
Population: PK Analysis Set: Includes all participants who have received at least 1 dose of the AMG 910 and have at least 1 PK sample collected. Participants with data available at each time point are included.
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Cohort 1: AMG 910 6.5 µg | Cohort 1b: AMG 910 6.5 µg | Cohort 2b: AMG 910 15 µg
Number analyzed (Participants) | 6 | 4 | 5
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 6 | 0 | 0
  Cycle 1 Day 1 | 3.78 [1.19 to 10.1] |  |
  Cycle 1 Day 3: number analyzed (Participants) | 5 | 0 | 0
  Cycle 1 Day 3 | 5.89 [2.02 to 17.2] |  |
  Cycle 1 Day 7: number analyzed (Participants) | 0 | 4 | 5
  Cycle 1 Day 7 |  | 2.91 [1.12 to 4.99] | 15.8 [1.47 to 30.2]
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 4 | 4
  Cycle 1 Day 8 | 2.92 [2.16 to 3.52] | 13.6 [1.63 to 47.6] | 22.3 [9.02 to 28.1]
  Cycle 1 Day 10: number analyzed (Participants) | 3 | 0 | 0
  Cycle 1 Day 10 | 3.62 [2.45 to 4.27] |  |
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 2 | 4
  Cycle 1 Day 15 | 1.82 [1.82 to 1.82] | 4.99 [1.35 to 8.62] | 10.5 [5.79 to 17.3]
  Cycle 1 Day 17: number analyzed (Participants) | 1 | 0 | 0
  Cycle 1 Day 17 | 2.17 [2.17 to 2.17] |  |
  Cycle 1 Day 22: number analyzed (Participants) | 1 | 0 | 0
  Cycle 1 Day 22 | 2.22 [2.22 to 2.22] |  |
  Cycle 1 Day 24: number analyzed (Participants) | 1 | 0 | 0
  Cycle 1 Day 24 | 2.38 [2.38 to 2.38] |  |

4. Secondary Outcome: Minimum Serum Concentration (Ctrough) of AMG 910
Description: Mean Ctrough values for the dosing intervals following short-term IV infusion (Cohort 1) and following extended IV infusions (Cohorts 1b and 2b) for Cycle 1 Week 1, and for short-term IV infusions in subsequent dosing intervals in Cycle 1 are presented. The timing of the PK sampling for Week 1 (Days 1-7) was based on hours after the start of infusion and from Day 8 onwards was based on hours after EOI. Due to the limited number of samples obtained and early termination of the study, PK data are summarized for Cycle 1 only.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Cohort 1: AMG 910 6.5 µg | Cohort 1b: AMG 910 6.5 µg | Cohort 2b: AMG 910 15 µg
Number analyzed (Participants) | 6 | 4 | 5
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 5 | 0 | 0
  Cycle 1 Day 1 | 0.952 [0.416 to 1.97] |  |
  Cycle 1 Day 3: number analyzed (Participants) | 4 | 0 | 0
  Cycle 1 Day 3 | 0.698 [0.450 to 1.21] |  |
  Cycle 1 Day 7: number analyzed (Participants) | 0 | 4 | 4
  Cycle 1 Day 7 |  | 0.813 [0.438 to 1.59] | 7.27 [2.24 to 11.0]
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 3 | 4
  Cycle 1 Day 8 | 1.48 [1.04 to 1.92] | 1.54 [0.316 to 3.40] | 3.70 [1.06 to 5.55]
  Cycle 1 Day 10: number analyzed (Participants) | 3 | 0 | 0
  Cycle 1 Day 10 | 0.979 [0.582 to 1.68] |  |
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 2 | 4
  Cycle 1 Day 15 | 0.836 [0.836 to 0.836] | 1.02 [0.00 to 2.03] | 2.54 [0.809 to 4.37]
  Cycle 1 Day 17: number analyzed (Participants) | 1 | 0 | 0
  Cycle 1 Day 17 | 0.664 [0.664 to 0.664] |  |
  Cycle 1 Day 22: number analyzed (Participants) | 1 | 0 | 0
  Cycle 1 Day 22 | 1.05 [1.05 to 1.05] |  |
  Cycle 1 Day 24: number analyzed (Participants) | 1 | 0 | 0
  Cycle 1 Day 24 | 0.540 [0.540 to 0.540] |  |

5. Secondary Outcome: Area Under the Concentration-time Curve (AUC) Over the Dosing Interval (AUC0_168hr)
Description: The timing of the PK sampling for Week 1 (Days 1-7) was based on hours after the start of infusion, and for Day 8 after EOI.
Time Frame: Cycle 1 Day 1 at pre-infusion, 1, 2, 4, 24, 48, 72, 96, 120 and 144 hr after infusion start and Cycle 1 Day 8 pre-infusion through 168 hr post-EOI
Population: PK Analysis Set: Includes all participants who have received at least 1 dose of the AMG 910 and have at least 1 PK sample collected. Participants with data available are included.
Measure: Mean (Standard Deviation); unit: hr•ng/mL
Arm/Group | Cohort 1: AMG 910 6.5 µg | Cohort 1b: AMG 910 6.5 µg | Cohort 2b: AMG 910 15 µg
Number analyzed (Participants) | 5 | 4 | 3
hr•ng/mL | 359 (262) | 251 (98.6) | 1710 (1160)

6. Secondary Outcome: Cohort 1 Only: Accumulation Ratio (AR) of AMG 910
Description: Calculated as AR = Cycle 1 Day 22 pre-infusion concentration/Cycle 1 Day 8 pre-infusion concentration.
Time Frame: Cycle 1 Day 8 pre-infusion and Cycle 1 Day 22 pre-infusion
Population: PK Analysis Set: Includes all participants who have received at least 1 dose of the AMG 910 and have at least 1 PK sample collected. Participants with data available at both time points are included.
Measure: Number; unit: ratio
Arm/Group | Cohort 1: AMG 910 6.5 µg
Number analyzed (Participants) | 1
ratio | 1.48

7. Secondary Outcome: Half-life (t1/2) of AMG 910
Description: Mean t1/2 values for the dosing intervals following short-term IV infusion (Cohort 1) and following extended IV infusions (Cohorts 1b and 2b) for Cycle 1 Week 1, and for short-term IV infusions in subsequent dosing intervals in Cycle 1 are presented. The timing of the PK sampling for Week 1 (Days 1-7) was based on hours after the start of infusion and from Day 8 onwards was based on hours after EOI. Due to the limited number of samples obtained and early termination of the study, PK data are summarized for Cycle 1 only.
Time Frame: Cycle 1: Days 1-7 at pre-infusion, 1, 2, 4, 24, 48, 72, 96, 120 and 144 hr; Days 8 and 10* at pre-infusion, EOI, 4 and 24 hr post-EOI (*=Cohort 1 only)
Population: as for outcome 3
Measure: Mean (Full Range); unit: hr
Arm/Group | Cohort 1: AMG 910 6.5 µg | Cohort 1b: AMG 910 6.5 µg | Cohort 2b: AMG 910 15 µg
Number analyzed (Participants) | 2 | 4 | 4
hr
  Cycle 1 Day 3: number analyzed (Participants) | 1 | 0 | 0
  Cycle 1 Day 3 | 47.4 [47.4 to 47.4] |  |
  Cycle 1 Day 7: number analyzed (Participants) | 0 | 2 | 0
  Cycle 1 Day 7 |  | 39.3 [33.5 to 45.1] |
  Cycle 1 Day 8: number analyzed (Participants) | 0 | 2 | 4
  Cycle 1 Day 8 |  | 63.2 [55.2 to 71.1] | 66.9 [60.0 to 74.0]
  Cycle 1 Day 10: number analyzed (Participants) | 1 | 0 | 0
  Cycle 1 Day 10 | 45.6 [45.6 to 45.6] |  |

8. Secondary Outcome: Number of Participants With an Objective Response (OR) Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Description: OR was defined as a best overall response (BOR) of complete response (CR) or partial response (PR) per RECIST v1.1:
  * CR: Disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have had a reduction in short axis to < 10 mm.
  * PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Non target lesions must be non-progressive Disease (non-PD).
Time Frame: Day 1 to end of study (EOS); maximum time on study was 18.76 months
Population: RECIST Evaluable Analysis Set: Included all participants that were enrolled and received at least 1 dose of AMG 910 with at least 1 tumor lesion that was measurable in contrast-enhanced computed tomography (CT) as defined by RECIST 1.1 at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: AMG 910 6.5 µg | Cohort 1b: AMG 910 6.5 µg | Cohort 2b: AMG 910 15 µg
Number analyzed (Participants) | 5 | 3 | 5
Participants | 0 | 0 | 0

9. Secondary Outcome: ORR Per Immune RECIST (iRECIST)
Description: ORR was defined as the incidence of a BOR of immune complete response (iCR) or immune partial response (iPR) per iRECIST:
  * iCR: Disappearance of all non-nodal target and non-target lesions and normalization of pathological lymph nodes (whether target or non-target) to <10 mm in short axis.
  * iPR: At least a 30% decrease in the sum of measures of target lesions, taking as reference the baseline target lesion sum.
  Data was not collected due to early termination of study, therefore data are not available.
Time Frame: Day 1 to EOS; maximum time on study was 18.76 months
Population: Data were not collected.
Arm/Group | Cohort 1: AMG 910 6.5 µg | Cohort 1b: AMG 910 6.5 µg | Cohort 2b: AMG 910 15 µg
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1
Description: As no participants experienced an objective response, data were not available.
Time Frame: Day 1 to EOS; maximum time on study was 18.76 months
Population: RECIST Evaluable Analysis Set: Included all participants that were enrolled and received at least 1 dose of AMG 910 with at least 1 tumor lesion that was measurable in contrast-enhanced CT as defined by RECIST 1.1 at baseline.
Arm/Group | Cohort 1: AMG 910 6.5 µg | Cohort 1b: AMG 910 6.5 µg | Cohort 2b: AMG 910 15 µg
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: DOR Per iRECIST
Description: Data was not collected due to early termination of study, therefore data are not available.
Time Frame: Day 1 to EOS; maximum time on study was 18.76 months
Population: Data were not collected.
Arm/Group | Cohort 1: AMG 910 6.5 µg | Cohort 1b: AMG 910 6.5 µg | Cohort 2b: AMG 910 15 µg
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Time to Progression Per RECIST 1.1
Description: Data was not collected due to early termination of study, therefore data are not available.
Time Frame: Day 1 to EOS; maximum time on study was 18.76 months
Population: Data were not collected.
Arm/Group | Cohort 1: AMG 910 6.5 µg | Cohort 1b: AMG 910 6.5 µg | Cohort 2b: AMG 910 15 µg
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Time to Progression Per iRECIST
Description: Data was not collected due to early termination of study, therefore data are not available.
Time Frame: Day 1 to EOS; maximum time on study was 18.76 months
Population: Data were not collected.
Arm/Group | Cohort 1: AMG 910 6.5 µg | Cohort 1b: AMG 910 6.5 µg | Cohort 2b: AMG 910 15 µg
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Progression-free Survival (PFS) Per RECIST 1.1
Description: Data was not collected due to limited follow up time due to study termination, therefore data are not available.
Time Frame: 6 months and 1 year
Population: Data were not collected.
Arm/Group | Cohort 1: AMG 910 6.5 µg | Cohort 1b: AMG 910 6.5 µg | Cohort 2b: AMG 910 15 µg
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: PFS Per iRECIST
Description: Data was not collected due to early termination of study, therefore data are not available.
Time Frame: 6 months and 1 year
Population: Data were not collected.
Arm/Group | Cohort 1: AMG 910 6.5 µg | Cohort 1b: AMG 910 6.5 µg | Cohort 2b: AMG 910 15 µg
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Overall Survival
Description: Data was not collected due to limited follow up time due to study termination, therefore data are not available.
Time Frame: 1 year and 2 years
Population: Data were not collected.
Arm/Group | Cohort 1: AMG 910 6.5 µg | Cohort 1b: AMG 910 6.5 µg | Cohort 2b: AMG 910 15 µg
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: For mortality reporting, "From enrollment until the end of study; median (min, max) time on study was 2.4 ( 0.43, 18.89) months". For AE reporting, "From first dose of study drug until 30 days after last dose; median (min, max) duration was 1.9 ( 0.43, 10.97) months".
Description: For all-cause mortality, time frame is from enrollment through end of study including long term follow-up. For SAE and non-serious AEs, time frame is treatment emergent.
Arm/Group | Cohort 1: AMG 910 6.5 µg | Cohort 1b: AMG 910 6.5 µg | Cohort 2b: AMG 910 15 µg
All-Cause Mortality (participants affected / at risk) | 4/6 | 3/4 | 2/5
Serious Adverse Events (participants affected / at risk) | 4/6 | 3/4 | 2/5
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: AMG 910 6.5 µg (N=6) | Cohort 1b: AMG 910 6.5 µg (N=4) | Cohort 2b: AMG 910 15 µg (N=5)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal stent stenosis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: AMG 910 6.5 µg (N=6) | Cohort 1b: AMG 910 6.5 µg (N=4) | Cohort 2b: AMG 910 15 µg (N=5)
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 2
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 1
Ascites (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Faecal vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 2 | 3
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1 | 2
Asthenia (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 3 | 1
Generalised oedema (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 2 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 2 | 2 | 2
COVID-19 (Infections and infestations) | 1 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Afferent loop syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Amylase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1
Lipase increased (Investigations) | 1 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Serum ferritin decreased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 1 | 0
Hypotension (Vascular disorders) | 2 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was discontinued due to a strategic decision to end clinical development for AMG 910 that was unrelated to safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT04260191/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT04260191/SAP_001.pdf